CLINICAL TRIAL: NCT01040533
Title: One-stage Laparoscopic Revision of Failed and/or Complicated Jejunoileal Bypass to Roux-en-Y Gastric Bypass
Brief Title: Laparoscopic Revision of Jejunoileal Bypass to Gastric Bypass
Acronym: JIB-to-RYGB
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Kelvin D Higa, MD; FACS; FASMBS; Professor of Surgery, University of California San Francisco, UCSF Fresno / ALSA Medical Group, Inc. Minimally Invasive Surgery Program
Other Study IDs: CMC IRB No. 2008085; U1111-1112-9885 (Other: World Health Organization, Universal Trial Number)
Record Dates: First submitted 2009-12-26; First posted 2009-12-29 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Clinically Severe Obesity; Metabolic Complications After Jejunoileal Bypass; Nutritional Complications After Jejunoileal Bypass; Obesity Recidivism; Inadequate Initial Weight Loss; Intestinal Malabsorptive Syndrome; Protein Malnutrition
Keywords: Failed jejunoileal bypass; Complicated jejunoileal bypass; Revision gastric bypass; Revisional surgery; Reoperations; Metabolic and nutritional complications
MeSH Terms: conditions — Kwashiorkor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Failed / complicated jejunoileal bypass

SUMMARY:
This study objectives are the following.

* To describe the updated clinical presentation, indications, and multidisciplinary medical management of patients with a failed and/or complicated jejunoileal bypass (JIB).
* To analyze the feasibility, safety, and efficacy of one-stage laparoscopic re-operative gastric bypass surgery for failed and/or complicated Jejunoileal bypass (JIB) for weight loss.
* To determine what factors or strategies are associated with a successful outcome. In particular, the completion of the surgery in one stage with a laparoscopic approach.

DETAILED DESCRIPTION:
The epidemic of overweight and obesity in the United States of America along with its comorbidities continues to expand. Bariatric surgery has demonstrated to be the most effective and sustained method to control severe obesity and its comorbidities. For instance, type 2 diabetes mellitus was completely resolved in 76.8 percent, systemic arterial hypertension was resolved in 61.7 percent, dyslipidemia improved in 70 percent, and obstructive sleep apnea hypopnea syndrome was resolved in 85.7 percent. Furthermore, bariatric surgery significantly increases life expectancy (89 percent) and decreases overall mortality (30 to 40 percent), particularly deaths from diabetes, heart disease, and cancer. Lastly, preliminary evidence about downstream savings associated with bariatric surgery offset the initial costs in 2 to 4 years8.

Since 1998, there has been a substantially progressive increase in bariatric surgery. In 2005, the American Society of Metabolic and Bariatric Surgery "ASMBS" reported that 81 percent of bariatric procedures were approached laparoscopically. 205,000 people, in 2007, had bariatric surgery in the United States from which approximately 80 percent of these were Gastric Bypass. Moreover, there is a mismatch between eligibility and receipt of bariatric surgery with just less than 1 percent of the eligible population being treated for morbid obesity through bariatric surgery. Along with the increasing number of elective primary weight loss procedures, up to 20 percent of post RYGB patients cannot sustain their weight loss beyond 2 to 3 years after the primary bariatric procedure. Thus, revisional surgery for poor weight loss and re-operations for technical or mechanical complications will rise in a parallel manner.

Regardless of being an effective treatment of morbid obesity, JIB was abandoned in the early 80s mostly because of its metabolic and nutritional complications. Multiple patients who underwent this procedure more than two decades ago are still alive. Close follow-up, in even asymptomatic patients, is necessary after JIB because they may present with nonreversible complications.

As with any bariatric procedure, weight regain, inadequate initial weight loss, and late complications or a combination of them are the most widely accepted indications to undergo revisional bariatric surgery. Specifically, the JIB related late complications can be arbitrarily categorized into "malabsorption and malnutrition" and "bacterial overgrowth syndrome". The former might present with steatorrhea, electrolyte (K, Ca, P, Mg) and acid base imbalance (hyperchloremic metabolic acidosis), liposoluble (A, D, E, K) and hydrosoluble (B1, B12 and Folate) vitamin deficiencies, and protein calorie malnutrition "PCM". "The bacterial overgrowth syndrome" causes a variety of complications such as gas bloat syndrome, foul smelling flatulence, recurrent migratory polyarthralgia and necrotizing skin lesions. Other late non metabolic complications related to the bypassed bowel include intussusception, pseudo-obstruction, and bypass enteropathy.

"PCM" is quickly and effectively treated by parenteral nutritional support. Diet optimization with consumption of high biological value protein (90 g per day) and a total calorie intake adjusted to ideal body weight might decrease the severity of the malabsorption syndrome and or prevent its recurrence.

Transitory resolution of most symptoms caused by the bacterial overgrowth syndrome is accomplished by the administration, in divided doses, of oral tetracycline (2.0 g per day), amoxicillin-clavulanate (1 to 1.7g per day), clindamycin (0.9 to 1.8 g per day), and metronidazole (1 to 1.5 g per day) among others. Rapid symptomatic improvement is observed, however, over time, organisms become resistant to the systemic absorption of antibiotics, ceasing the benefit of this therapy. In addition, side effects including superinfections such as pseudomembranous colitis might present. Local instillation of antibiotic through an intestinal indwelling catheter placed in the excluded bowel limb has been described.

When the JIB related complications present as intractable, severe or recurrent, surgical intervention is required. Liver, either acute liver failure or cirrhosis, (secondary to "PCM" and bacterial overgrowth syndrome) and kidney, either tubulointerstitial nephropathy or renoureteral lithiasis, (secondary to enteric hyperoxaluria and volume depletion) dysfunction are the most frequently described complications leading to death. However, after end stage liver (cirrhosis) and renal diseases are established, good judgment is needed to assess the risk benefit algorithm for operative intervention, as these conditions are irreversible.

In the United States, the most popular type of intestinal bypass performed was the so called "14 plus 4" with an end to side jejunoileostomy, a 14 inches biliopancreatic limb with a 4 inches common channel. Because of poor weight loss, some surgeons used to performed an end to end jejunoileostomy avoiding chyme to reflux into the defunctionalized limb; Through an ileocolostomy, the defunctionalized jejunoileal limb was drained into the cecum or sigmoid colon.

Open reversal or conversion to gastric bypass has been shown to be effective procedures with defined complications. Since the 60s Payne, DeWind and Commons had already demonstrated that takedown and restitution of the gastrointestinal continuity is an effective strategy to solve the metabolic complications. However, relapse of obesity along with its comorbidities is the rule.

Series from the 70s and 80s suggested that one stage open revision of JIB to gastric bypass was feasible and safe. However, most of these revisions were performed a couple of years after the original bariatric surgery with a completely different configuration (non divided horizontal pouch with a loop gastrojejunostomy) from how modern RYGB is performed in these days. Hence, outcome analysis of those series is not transferable in today context.

Because of the long interval time between the JIB and the revision surgery, bowel adaptation is maximal causing a marked discrepancy in the lumen diameter and bowel thickness between the functional and defunctionalized bowel segments. Thus, different approaches have been described in the literature to deal with more extensive intestinal changes..

Based on Cannova et al. report in which described the placement of an intestinal indwelling catheter in the excluded bowel limb, Dallal et al. with a minimally invasive approach established enteral nutritional support in the defunctionalized bowel limb, to revert its atrophy. After a three month period with extensive counseling to undergo conversion to a RYGB, the patient decided just to be reversed.

Another staged option for revising the JIB is as follows. Initially, the JIB is dismantled and the normal gastrointestinal continuity restored. After the initially bypassed and atrophied small bowel regains its function and the bowel atrophy is partially overturned, the second stage (weight loss procedure) is performed, so weight loss can be maintained or achieved.

The two accepted revisionary procedures described in the literature for failed JIB are mainly adjustable gastric banding (AGB) and gastric bypass. In 2000, O'Brien et al. reported a series of 50 revisions to adjustable gastric banding. As the primary bariatric procedure, two patients had a JIB. A one stage open revision was performed without providing specific subset outcome analysis.

In 1993, Behrns et al. reported the outcome analysis of 61 open assorted revision surgeries from which 14 had a JIB. The indication for this subgroup was due to severe metabolic complications with a pre-revisional mean BMI of 34.2 kilograms per squared meter. Nine patients were revised to VBG and five patients to a non-divided, vertical RYGB. The percent excess weight loss for this five patients was 49.5 percent (overall follow-up was 23 months) with a 67 percent dissatisfaction rate of their new lifestyle because of the change in eating patterns caused by switching from a full size meal to a restricted diet.

In 1996, Owens et al. reported the open surgical revision of 75 patients from which 23 patients had a JIB as their primary procedure. Specific subgroup analysis was not provided. In 2005, khaitan et al. reported 37 patients who underwent 39 bariatric revisions, either open or laparoscopic. Originally, five had a JI bypass from which two were initially approached laparoscopically. However, specific subgroup analysis was not provided.

In summary, there are just two manuscripts reporting cases of attempted laparoscopic conversion of JIB to RYGB with its modern anatomical construction. However, a one stage procedure has not been achieved up to date. Therefore, no outcomes with this approach have been documented as well. With this study, we will advance our knowledge about revision bariatric surgery and report excellent outcomes after conversion from a completely malabsorptive procedure to a mostly restrictive weight loss procedure, the gastric bypass and although JIB was abandoned long time ago, there are still living patients with this procedure and bariatric surgeons need to be aware of side effects and minimally invasive strategies for the management of these highly complex patients.

ELIGIBILITY:
Inclusion Criteria:

* Met NIH criteria for weight loss surgery with poor weight loss after JIB
* Intractable, severe and/or recurrent JIB-related late complications after optimized medical management
* Laparoscopic approach for primary revisional bariatric surgery

Exclusion Criteria:

* Any other type of revisional bariatric procedure
* Open approach for revision surgery
* missing records and/or unreachable patients with scant information for analysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent laparoscopic revision of JIB to Roux-en-Y gastric bypass (RYGB) for poor weight loss or JIB-related late complications were analyzed. Failed or JIB-related late complications, mostly metabolic, were considered for surgical intervention after optimized medical multidisciplinary management
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Morbidity and mortality | throughout follow-up
Weight loss expressed as Body Mass Index and Percentage excess weight loss | throughout follow-up
Remission or improvement of symptoms and JIB-related complications | throughout follow-up
Remission or improvement of other comorbidities | throughout follow-up

SECONDARY OUTCOMES:
Operative time | transoperatively
conversion to open approach | transoperatively
Hospital stay | same hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Tercero, MD, Study Director — Research Associate, University of California San Francisco; Kelvin D Higa, MD, Principal Investigator — Professor of Surgery, University of California San Francisco
Locations (1):
- UCSF Fresno Center for Medical Education and Research, Department of Surgery, Fresno, California, United States

REFERENCES:
- [Background] Higa KD, Boone KB, Ho T, Davies OG. Laparoscopic Roux-en-Y gastric bypass for morbid obesity: technique and preliminary results of our first 400 patients. Arch Surg. 2000 Sep;135(9):1029-33; discussion 1033-4. doi: 10.1001/archsurg.135.9.1029. PMID 10982506
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] McTigue KM, Harris R, Hemphill B, Lux L, Sutton S, Bunton AJ, Lohr KN. Screening and interventions for obesity in adults: summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2003 Dec 2;139(11):933-49. doi: 10.7326/0003-4819-139-11-200312020-00013. PMID 14644897
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004 Sep;240(3):416-23; discussion 423-4. doi: 10.1097/01.sla.0000137343.63376.19. PMID 15319713
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Cremieux PY, Buchwald H, Shikora SA, Ghosh A, Yang HE, Buessing M. A study on the economic impact of bariatric surgery. Am J Manag Care. 2008 Sep;14(9):589-96. PMID 18778174
- [Background] Santry HP, Gillen DL, Lauderdale DS. Trends in bariatric surgical procedures. JAMA. 2005 Oct 19;294(15):1909-17. doi: 10.1001/jama.294.15.1909. PMID 16234497
- [Background] Flum DR, Khan TV, Dellinger EP. Toward the rational and equitable use of bariatric surgery. JAMA. 2007 Sep 26;298(12):1442-4. doi: 10.1001/jama.298.12.1442. No abstract available. PMID 17895461
- [Background] Meguid MM, Glade MJ, Middleton FA. Weight regain after Roux-en-Y: a significant 20% complication related to PYY. Nutrition. 2008 Sep;24(9):832-42. doi: 10.1016/j.nut.2008.06.027. PMID 18725080
- [Background] Nguyen NT. Reoperations and revisions in bariatric surgery. Surg Endosc. 2007 Nov;21(11):1907-8. doi: 10.1007/s00464-007-9572-6. Epub 2007 Sep 8. No abstract available. PMID 17828427
- [Background] Bradley JE, Brown RO, Luther RW. Multiple nutritional deficiencies and metabolic complications 20 years after jejunoileal bypass surgery. JPEN J Parenter Enteral Nutr. 1987 Sep-Oct;11(5):494-8. doi: 10.1177/0148607187011005494. PMID 3116298
- [Background] Gasbarrini A, Lauritano EC, Gabrielli M, Scarpellini E, Lupascu A, Ojetti V, Gasbarrini G. Small intestinal bacterial overgrowth: diagnosis and treatment. Dig Dis. 2007;25(3):237-40. doi: 10.1159/000103892. PMID 17827947
- [Background] Wands JR, LaMont JT, Mann E, Isselbacher KJ. Arthritis associated with intestinal-bypass procedure for morbid obesity. Complement activation and characterization of circulating cryoproteins. N Engl J Med. 1976 Jan 15;294(3):121-4. doi: 10.1056/NEJM197601152940301. PMID 1105187
- [Background] Cannova JV, Krummen DM, Schreiber H, Schaefer IK. An approach to the treatment of recurring polyarthralgia after jejunoileal bypass. Obes Surg. 1997 Jun;7(3):215-7; discussion 218-9. doi: 10.1381/096089297765555773. PMID 9730552
- [Background] Buckwalter JA, Herbst CA Jr. Reversal of jejunoileal bypass. Surg Gynecol Obstet. 1984 Oct;159(4):348-52. PMID 6484791
- [Background] Pessa M, Robertson J, Woodward ER. Surgical management of the failed jejunoileal bypass. Am J Surg. 1986 Mar;151(3):364-7. doi: 10.1016/0002-9610(86)90469-1. PMID 3953955
- [Background] Tapper D, Hunt TK, Allen RC, Campbell J. Conversion of jejunoileal bypass to gastric bypass to maintain weight loss. Surg Gynecol Obstet. 1978 Sep;147(3):353-7. PMID 684586
- [Background] LaFave JW, Alden JF. Gastric bypass in the operative revision of the failed jejunoileal bypass. Arch Surg. 1979 Apr;114(4):438-44. doi: 10.1001/archsurg.1979.01370280092013. PMID 435057
- [Background] Griffen WO Jr, Hostetter JM, Bell RM, Bivins BA, Bannon C. Experiences with conversion of jejunoileal bypass to gastric bypass: its use for maintenance of weight loss. Arch Surg. 1981 Mar;116(3):320-4. doi: 10.1001/archsurg.1981.01380150048013. PMID 7469774
- [Background] Charuzi I, Grizim D, Peiser J, Solomon H, Ovnat A. Simultaneous replacement of a failed jejunoileal bypass with a gastric bypass. Isr J Med Sci. 1984 Dec;20(12):1183-5. PMID 6519951
- [Background] Ackerman NB. Metabolic consequences from conversion of jejunoileal bypass to gastric bypass. Ann Surg. 1982 Nov;196(5):553-9. doi: 10.1097/00000658-198211000-00007. PMID 7125740
- [Background] Dallal RM, Akhondzadeh M. Minimally invasive management of complications from jejunoileal bypass. Surg Obes Relat Dis. 2006 Mar-Apr;2(2):226-7. doi: 10.1016/j.soard.2006.01.006. Epub 2006 Feb 28. No abstract available. PMID 16925349
- [Background] O'Brien P, Brown W, Dixon J. Revisional surgery for morbid obesity--conversion to the Lap-Band system. Obes Surg. 2000 Dec;10(6):557-63. doi: 10.1381/096089200321594174. PMID 11175966
- [Background] Behrns KE, Smith CD, Kelly KA, Sarr MG. Reoperative bariatric surgery. Lessons learned to improve patient selection and results. Ann Surg. 1993 Nov;218(5):646-53. doi: 10.1097/00000658-199321850-00010. PMID 8239779
- [Background] Khaitan L, Van Sickle K, Gonzalez R, Lin E, Ramshaw B, Smith CD. Laparoscopic revision of bariatric procedures: is it feasible? Am Surg. 2005 Jan;71(1):6-10; discussion 10-2. PMID 15757050
- [Background] Raftopoulos I, Courcoulas AP. Revision of jejunoileal bypass to Roux-en-Y gastric bypass: technical considerations and outcomes from 2 cases. Surg Obes Relat Dis. 2008 Mar-Apr;4(2):198-201. doi: 10.1016/j.soard.2007.10.009. Epub 2007 Dec 11. No abstract available. PMID 18065288
- See also: "Click here for more information about the department sponsor´s web site" — http://www.fresno.ucsf.edu/surgery/